CLINICAL TRIAL: NCT06935591
Title: Artificial Intelligence Mapping and Ablation of Non-Pulmonary Vein Electrical Drivers of AF Study
Acronym: IMPRoVED-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vektor Medical (Industry)
Collaborators: Veranex Switzerland SA (Industry); Veranex (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-VM-1001
Record Dates: First submitted 2025-04-08; First posted 2025-04-20 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Pulmonary Vein Isolation; Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a post-market, prospective, multi-center, two-arm randomized-controlled clinical study. Subjects will be randomized in a 1:1 ratio into two arms: a treatment arm (use of vMap® system in addition to pulmonary vein isolation [vMap®+PVI]) and a control arm (PVI alone). The study is designed to compare clinical outcomes following use of an FDA-cleared/commercially available forward-solution computational 12-lead ECG mapping system (vMap®) for identifying/mapping for subjects who are indicated to undergo ablation procedures for persistent and recurrent AF in accordance with standard of care practices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- vMap®+PVI (Experimental): Subjects in this arm will be treated with the use of the vMap® system in addition to pulmonary vein isolation.
  Interventions: Device: vMap® + Pulmonary Vein Isolation
- PVI Alone (Active Comparator): Subjects in this arm will be treated with pulmonary vein isolation alone.
  Interventions: Procedure: Pulmonary Vein Isolation

INTERVENTIONS:
Procedure: Pulmonary Vein Isolation — Subjects will receive treatment for Atrial Fibrillation with Pulmonary Vein Isolation per standard of care.
  Arms: PVI Alone
Device: vMap® + Pulmonary Vein Isolation — Subjects will receive treatment for Atrial Fibrillation with the use of the vMap® system and Pulmonary Vein Isolation.
  Arms: vMap®+PVI

SUMMARY:
The goal of this clinical trial is to compare the use of the Vektor Computational ECG Mapping System (vMap®) with pulmonary vein isolation (PVI), to using PVI alone, to treat Atrial Fibrillation (AF) in adults.

Participants will have a 50/50 or 1 out of 2 chance of being placed in the treatment or control arm. The control arm of the study involves PVI alone for ablation procedure(s). The treatment arm involves the use of vMap mapping in addition to PVI to plan ablation procedure(s).

DETAILED DESCRIPTION:
This is a post-market, prospective, multi-center, two-arm randomized-controlled clinical study. Subjects will be randomized in a 1:1 ratio into two arms: a treatment arm (use of vMap® system in addition to pulmonary vein isolation [vMap®+PVI]) and a control arm (PVI alone). The study is designed to compare clinical outcomes following use of an FDA-cleared/commercially available forward-solution computational 12-lead ECG mapping system (vMap®) for identifying/mapping for subjects who are indicated to undergo ablation procedures for persistent and recurrent AF in accordance with standard of care practices.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with persistent (not longstanding) AF or recurrent AF, as defined for this study.
2. Subject has a recent 12-lead electrogram data of AF (including baseline, pacing and clinical arrhythmia) recorded on the electrogram recording system (e.g., Bard, Boston-Scientific, St. Paul, MN or Prucka, GE Medical) or standalone ECG system (e.g., GE Muse, Minnesota, or CardioCard (Nasiff, NY) in digitized format.
3. The following data elements can be abstracted from the patient medical records or confirmed and documented prior to the scheduled procedure (to be inputted in vMap®):

   * Atrial fibrillation type
   * Atrial characteristics: geometry (normal, left and/or right atrial enlargement), Utah classification, prior ablation modality (e.g., radiofrequency, cryoablation, pulsed field ablation), prior ablation lesion location(s).
4. Subject is ≥ 22 years of age at time of enrollment/consent.
5. Subject is indicated to undergo an ablation procedure at the medical discretion of the Investigator.
6. Subject is able and willing to comply with the protocol requirements, has been informed of the nature of the study,

Exclusion Criteria:

1. Subjects with arrhythmias other than persistent or recurring AF as defined for this study, including long-standing persistent atrial fibrillation (persistent AF lasting ≥ 1 year from diagnosis).
2. Inability to obtain ECG prior to or during the clinical ablation procedure; or unacceptable ECG data quality such as low ECG signal-to-noise ratio or lack of ECG data in one or more leads.
3. Subjects who are participating in another clinical investigation with an investigational drug or device at the time of enrollment or planned participation at any time during this clinical investigation.
4. Subjects who have a known or suspected medical condition that, in the opinion of the Investigator, may put the subject at risk for participation in this clinical investigation.
5. Subjects who are pregnant as confirmed by the institution's standard pre-surgery practice.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from AF | 12 months post procedure
  The achievement of freedom from AF for subjects on or off antiarrhythmic drug (AAD) therapy at 12 months.

SECONDARY OUTCOMES:
Freedom from AF and AT | 12 months post procedure
  Freedom from both AF and AT for subjects on and off antiarrhythmic drug (AAD) therapy at 12 months.
Total Procedure Time | Interventional Procedure
  Defined as the time from completing intravascular access (successful placement of all vascular sheaths) to initiating hemostasis (time at which the first vascular sheath is removed from the subject).
Total vMap® Mapping Time | Interventional Procedure
  Defined as time from entering the ECG and patient characteristics into the vMap® and ending with display of the 3-dimensional mapping result, prior to delivery of the first ablation.
AF Burden | 12 months post procedure
  AF burden as a proportion of time before versus after the ablation procedure, excluding the 'blanking period'.
Spontaneous AF Termination | Interventional Procedure
  Proportion of subjects whose AF terminated spontaneously upon and after the first ablation lesion and before achieving hemostasis without cardioversion.
Total Fluoroscopy Dose | Interventional Procedure
  Defined as the cumulative dose-area product (DAP) for the procedure.

OTHER OUTCOMES:
Total Fluorscopy Time | 1Interventional Procedure
  Defined as the total time of fluoroscopy during procedure

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - Baptist Health Jacksonville, Jacksonville, Florida
  - USF Health, Tampa, Florida
  - Indiana University, Indianapolis, Indiana
  - Baptist Health Lexignton, Lexington, Kentucky
  - Westchester Medical Center, Valhalla, New York
  - OhioHealth, Columbus, Ohio
  - Penn Presbyterian, Philadelphia, Pennsylvania
- Catharina Ziekenhuis, Eindhoven, North Brabant, Netherlands